CLINICAL TRIAL: NCT01579370
Title: A Four-arm Prospective, Multicenter Study to Assess the Efficacy, Effectiveness, and Feasibility of Enhanced Terminal Room Disinfection With Chlorine and UV Light Using Clinical and Microbiologic Outcomes
Brief Title: Effectiveness of Enhanced Terminal Room Disinfection to Prevent Healthcare-associated Infections (HAIs)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: Pro00032718; 1U54CK000164-01 (NIH)
Record Dates: First submitted 2012-04-05; First posted 2012-04-18 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Multidrug Resistant Organisms; Healthcare Associated Infections
Keywords: healthcare associated infections; multidrug resistant organisms; methicillin resistant staphylococcus aureus; vancomycin resistant enterococcus; clostridium difficile; acinetobacter
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Quaternary ammonium (Active Comparator): Rooms will be terminally cleaned using quaternary ammonium-containing compounds, the reference standard for hospital cleaning in US hospitals.
  Interventions: Other: Quaternary ammonium
- Bleach (Experimental): Rooms will be terminally cleaned using bleach-containing products.
  Interventions: Other: Bleach
- Quaternary ammonium and UV-C light (Experimental): Rooms will be terminally cleaned with quaternary ammonium-containing solutions followed by irradiation by a UV-C light emitting device.
  Interventions: Other: Quaternary ammonium and UV-C light
- Bleach and UV-C light (Experimental): Rooms will be terminally cleaned with bleach-containing solutions followed by irradiation by a UV-C light emitting device.
  Interventions: Other: Bleach and UV-C light

INTERVENTIONS:
Other: Quaternary ammonium — Rooms from which a patient with a target organisms has been discharged (ie, a "seed" room) will be cleaned using quaternary-ammonium containing solutions. Room cleaning will proceed following standard cleaning protocols established at each study hospital.
  Arms: Quaternary ammonium
Other: Bleach — Rooms from which a patient with a target organisms has been discharged (ie, a "seed" room) will be cleaned using bleach containing solutions. Room cleaning will proceed following standard cleaning protocols established at each study hospital.
  Arms: Bleach
Other: Quaternary ammonium and UV-C light — Rooms from which a patient with a target organisms has been discharged (ie, a "seed" room) will be cleaned using quaternary-ammonium containing solutions. Room cleaning will proceed following standard cleaning protocols established at each study hospital. Then, the UV-C light-emitting device will be brought to the room to irradiate the room until 12,000 uWs/cm2 (for vegetative bacteria) or 22,000 uWs/cm2 (for C. difficile) has been delivered to entire room.
  Arms: Quaternary ammonium and UV-C light
Other: Bleach and UV-C light — Rooms from which a patient with a target organisms has been discharged (ie, a "seed" room) will be cleaned using bleach containing solutions. Room cleaning will proceed following standard cleaning protocols established at each study hospital. Then, the UV-C light-emitting device will be brought to the room to irradiate the room until 12,000 uWs/cm2 (for vegetative bacteria) or 22,000 uWs/cm2 (for C. difficile) has been delivered to entire room.
  Arms: Bleach and UV-C light

SUMMARY:
Enhanced terminal room disinfection is a novel, promising, but still unproven strategy for the prevention of healthcare-associated infections (HAIs) due to selected multidrug-resistant (MDR) bacterial pathogens. The investigators will perform a large prospective, multicenter study enhanced terminal room disinfection to 1) determine the efficacy and feasibility of enhanced terminal room disinfection strategies to prevent HAIs and 2) determine the impact of environmental contamination on acquisition of MDR-pathogens among hospitalized patients.

DETAILED DESCRIPTION:
Meticulous and consistent use of hand hygiene before and after patient care remains the cornerstone of infection prevention in all health care settings. However, clean hands are not sufficient to prevent all healthcare-associated infections (HAIs), as 1) hands of healthcare workers easily become contaminated from contact with contaminated environmental surfaces in patient rooms after appropriate hand hygiene has been performed and before direct patient care and 2) direct contact by patients with preexisting contaminated environmental surfaces in their hospital rooms can lead to colonization or infection. Thus, novel strategies are needed to prevent HAIs, particularly those caused by multidrug-resistant (MDR) pathogens that persist in the environment such as methicillin-resistant Staphylococcus aureus (MRSA), vancomycin-resistant Enterococci (VRE), Clostridium difficile, and Acinetobacter.

Enhanced environmental disinfection methods may lead to reduced risk of exposure to or acquisition of HAIs and MDR-pathogens and overcome a critical issue facing healthcare today - hospitals rooms are often poorly cleaned and disinfected. Enhanced terminal room disinfection strategies using bleach and/or UV-C emitting devices have been investigated only in experimental conditions; the efficacy, effectiveness, and feasibility of enhanced terminal room disinfection to prevent HAIs are unknown. Thus, the scientific evidence for such interventions currently is insufficient for their inclusion in evidence-based guidelines.

This study will investigate the hypothesis that enhanced terminal room disinfection protocols (using chlorine-based cleaning agents with or without UV-C light-emitting devices) will decrease the overall risk of HAIs in the hospital and, more specifically, in subsequent patients who are cared for in the same room. This prospective investigation will employ a crossover design utilizing four room cleaning/disinfection protocols in 9 hospitals, including 2 tertiary care, 1 VA, and 6 community hospitals. Phase T2 data from this study will be useful in assessing the clinical efficacy and feasibility of individual disinfection strategies. Thus, the goals of the investigators proposed research are to 1) determine the efficacy and feasibility of enhanced terminal room disinfection strategies to prevent HAIs and 2) determine the impact of environmental contamination on acquisition of MDR-pathogens among hospitalized patients.

ELIGIBILITY:
Inclusion Criteria:

* Any seed room (ie., room from which a patient with one of the target organisms has been transferred or discharged)

Exclusion Criteria:

* None, intervention is at level of the room, not the patient
* Patient outcomes will be excluded if clinical cultures are obtained within 48 hours of admission to the room of interest.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21395 (Actual)
Dates: Start 2012-04; Primary Completion 2014-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Clinical incidence rate of four target organisms among patients admitted to a study room | 90 days
  Patients will be monitored for clinical cultures that grow one of four target organisms (MRSA, VRE, C. difficile, and MDR-Acinetobacter) following admission to a "seed" room. Cultures for vegetative bacteria (MRSA, VRE, Acinetobacter) will be included if obtained within 90 days of discharge from a seed room; cultures for C. difficile will be included if they are obtained within 28 days of discharge from a seed room.
Clinical incidence rate of C. difficile among patients admitted to a study room | 28 days
  Patients will be monitored for clinical cultures that grow C. difficile following admission to a "seed" room.

SECONDARY OUTCOMES:
Clinical incidence rate of target vegetative bacteria (MRSA, VRE, Acinetobacter) among patients admitted to a seed room. | 90 days
  Patients will be monitored for clinical cultures that grow one of three target vegetative organisms (MRSA, VRE, and MDR-Acinetobacter) following admission to a "seed" room.
Clinical incidence rate of target organisms among all patients admitted to the hospital | 90 days
  All hospitalized patients will be monitored for clinical cultures that grow one of four target organisms (MRSA, VRE, C. difficile, and MDR-Acinetobacter) regardless of exposure to seed room.
Clinical incidence rate of MRSA among all patients admitted to the hospital | 90 days
  All hospitalized patients will be monitored for clinical cultures that grow MRSA regardless of exposure to seed room.
Clinical incidence rate of VRE among all patients admitted to the hospital | 90 days
  All hospitalized patients will be monitored for clinical cultures that grow VRE regardless of exposure to seed room.
Clinical incidence rate of MDR-Acinetobacter among all patients admitted to the hospital | 90 days
  All hospitalized patients will be monitored for clinical cultures that grow MDR-Acinetobacter regardless of exposure to seed room.
Clinical incidence rate of C. difficile among all patients admitted to the hospital | 28 days
  All hospitalized patients will be monitored for clinical cultures that grow C. difficile regardless of exposure to seed room.
Incidence rate of healthcare-associated infections caused by target bacteria (MRSA, VRE, C. difficile, and MDR-Acinetobacter) among patients admitted to a seed room. | Patients will be followed an average of 30 days
  Patients will be monitored for HAIs due to one of four target organisms (MRSA, VRE, C. difficile, and MDR-Acinetobacter) following admission to a "seed" room. NHSN definitions for HAIs will be used.
Incidence rate of healthcare-associated infections caused by MRSA among patients admitted to a seed room. | Patients will be followed an average of 30 days
  Patients will be monitored for HAIs due to MRSA following admission to a "seed" room. NHSN definitions for HAIs will be used.
Incidence rate of healthcare-associated infections caused by VRE among patients admitted to a seed room. | Patients will be followed an average of 30 days
  Patients will be monitored for HAIs due to VRE following admission to a "seed" room. NHSN definitions for HAIs will be used.
Incidence rate of healthcare-associated infections caused by MDR-Acinetobacter among patients admitted to a seed room. | Patients will be followed an average of 30 days
  Patients will be monitored for HAIs due to MDR-Acinetobacter following admission to a "seed" room. NHSN definitions for HAIs will be used.
Incidence rate of healthcare-associated infections caused by MDR-Acinetobacter among all hospitalized patients. | Patients will be followed an average of 30 days
  Patients will be monitored for HAIs due to MDR-Acinetobacter, regardless of exposure to seed room. NHSN definitions for HAIs will be used.
Incidence rate of healthcare-associated infections caused by MRSA among all hospitalized patients. | Patients will be followed an average of 30 days
  Patients will be monitored for HAIs due to MRSA, regardless of exposure to seed room. NHSN definitions for HAIs will be used.
Incidence rate of healthcare-associated infections caused by VRE among all hospitalized patients. | Patients will be followed an average of 30 days
  Patients will be monitored for HAIs due to VRE, regardless of exposure to seed room. NHSN definitions for HAIs will be used.
Incidence rate of healthcare-associated infections caused by target vegetative bacteria (MRSA, VRE, MDR-Acinetobacter) among all hospitalized patients. | Patients will be followed an average of 30 days
  Patients will be monitored for HAIs due to MRSA, VRE, and MDR-Acinetobacter regardless of exposure to seed room. NHSN definitions for HAIs will be used.
Missed Opportunities | each study period (6 months)
  Use of UV-C emitting devices will be monitored and "missed opportunities" (ie, UV-C emitter should have been used per protocol and was not) will be tracked and summarized. This proportion will be calculated for each study arm, each of which lasts 6 months. The "quaternary ammonium" (and no UV-C light) arm will be considered the reference group.
Time on Diversion | Each study period (6 months)
  Hospital data will be gathered to determine if use of UV-C emitting devices leads to downstream effects on hospital process. The proportion will be calculated as the average number of days on diversion per month for each study period. This proportion will be calculated for each study arm, each of which lasts 6 months. The "quaternary ammonium" (and no UV-C light) will be considered the reference group.
Room Turnover Time | Each study period (6 months)
  Room cleaning process will be monitored and tracked. We will obtain start and stop times for terminal room cleaning to determine if use of UV-C light emitting devices leads to additional time for room turnover. Average times will be calculated for each study arm, each of which lasts 6 months. The "quaternary ammonium" (and no UV-C light) arm will be considered the reference group.
ED to floor wait time | Each study period (6 months)
  Hospital data will be gathered to determine if use of UV-C emitting devices leads to downstream effects on hospital process. Average times will be calculated for each study arm, each of which lasts 6 months. The "quaternary ammonium" (and no UV-C light) arm will be considered the reference group.
Clinical incidence of MRSA, VRE, C. difficile, and MDR-Acinetobacter during UV-C light versus No UV-C light | 12 months (2 6-month study arms combined)
  The clinical incidence rate of MRSA, VRE, C. difficile, and MDR-Acinetobacter will be calculated for the two 6-month study arms (12 months total) during which UV-C light is used for terminal room disinfection (regardless of which chemical is used) and compared to the two 6-month study arms (12 months total) during which UV-C light is not used for terminal room disinfection.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Sexton, MD, Principal Investigator — Duke University
Locations (9):
- United States (9):
  - Alamance Regional Medical Center, Burlington, North Carolina
  - University of North Carolina Hospitals, Chapel Hill, North Carolina
  - Durham Regional Hospital, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Durham VA Medical Center, Durham, North Carolina
  - High Point Regional Health System, High Point, North Carolina
  - Rex Healthcare, Raleigh, North Carolina
  - Duke Raleigh Hospital, Raleigh, North Carolina
  - Chesapeake Regional Medical Center, Chesapeake, Virginia

REFERENCES:
- [Derived] Rutala WA, Kanamori H, Gergen MF, Knelson LP, Sickbert-Bennett EE, Chen LF, Anderson DJ, Sexton DJ, Weber DJ; and the CDC Prevention Epicenters Program. Enhanced disinfection leads to reduction of microbial contamination and a decrease in patient colonization and infection. Infect Control Hosp Epidemiol. 2018 Sep;39(9):1118-1121. doi: 10.1017/ice.2018.165. Epub 2018 Jul 31. PMID 30060770
- [Derived] Anderson DJ, Moehring RW, Weber DJ, Lewis SS, Chen LF, Schwab JC, Becherer P, Blocker M, Triplett PF, Knelson LP, Lokhnygina Y, Rutala WA, Sexton DJ; CDC Prevention Epicenters Program. Effectiveness of targeted enhanced terminal room disinfection on hospital-wide acquisition and infection with multidrug-resistant organisms and Clostridium difficile: a secondary analysis of a multicentre cluster randomised controlled trial with crossover design (BETR Disinfection). Lancet Infect Dis. 2018 Aug;18(8):845-853. doi: 10.1016/S1473-3099(18)30278-0. Epub 2018 Jun 4. PMID 29880301
- [Derived] Anderson DJ, Knelson LP, Moehring RW, Lewis SS, Weber DJ, Chen LF, Triplett PF, Blocker M, Cooney RM, Schwab JC, Lokhnygina Y, Rutala WA, Sexton DJ; CDC Prevention Epicenters Program. Implementation Lessons Learned From the Benefits of Enhanced Terminal Room (BETR) Disinfection Study: Process and Perceptions of Enhanced Disinfection with Ultraviolet Disinfection Devices. Infect Control Hosp Epidemiol. 2018 Feb;39(2):157-163. doi: 10.1017/ice.2017.268. Epub 2018 Jan 14. PMID 29331170
- [Derived] Anderson DJ, Chen LF, Weber DJ, Moehring RW, Lewis SS, Triplett PF, Blocker M, Becherer P, Schwab JC, Knelson LP, Lokhnygina Y, Rutala WA, Kanamori H, Gergen MF, Sexton DJ; CDC Prevention Epicenters Program. Enhanced terminal room disinfection and acquisition and infection caused by multidrug-resistant organisms and Clostridium difficile (the Benefits of Enhanced Terminal Room Disinfection study): a cluster-randomised, multicentre, crossover study. Lancet. 2017 Feb 25;389(10071):805-814. doi: 10.1016/S0140-6736(16)31588-4. Epub 2017 Jan 17. PMID 28104287